CLINICAL TRIAL: NCT01657136
Title: Comparison of Ivabradine and Beta-blockers Administration in the Treatment of Inappropriate Sinus Tachycardia
Brief Title: Ivabradine Versus Beta-blockers in the Treatment of Inappropriate Sinus Tachycardia
Acronym: CIBIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Leonardo Calo, Director of clinical arrhythmology and cardiac electrophysiology department, Policlinico Casilino ASL RMB
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Casilino0001; 0001
Record Dates: First submitted 2012-07-30; First posted 2012-08-06 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Inappropriate Sinus Tachycardia
Keywords: Inappropriate sinus tachycardia; ivabradine; beta blockers
MeSH Terms: interventions — Ivabradine; Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivabradine (Active Comparator): Ivabradine will be initiated at a dose of 5 mg twice daily. Dosage should be augmented up to 7.5 mg twice daily in case of symptoms persistence and/or HR > 85 bpm at rest ECG and eventually lowered up to 2.5 mg twice daily in the presence of side effects (phosphenes, diplopia and symptomatic bradycardia).
  Interventions: Drug: Ivabradine
- Beta blocker (Bisoprololo) (Active Comparator): Bisoprololo will be initiated at a single dose of 5 mg daily. Dosage should be augmented up to 10 mg single dose daily in case of symptoms persistence and/or HR > 85 bpm at rest ECG and eventually lowered up to 2,5 mg single dose daily in the presence of side effects (symptomatic bradycardia, hypotension).
  Interventions: Drug: Beta blocker

INTERVENTIONS:
Drug: Ivabradine — comparison of different drugs
  Arms: Ivabradine
Drug: Beta blocker — comparison of different drugs
  Arms: Beta blocker (Bisoprololo)

SUMMARY:
The aim of this study is to prospectively compare the effectiveness and safety of ivabradine and beta-blockers in the treatment of inappropriate sinus tachycardia.

DETAILED DESCRIPTION:
Inappropriate sinus tachycardia (IST) is a non-paroxysmal arrhythmia, characterized by a persistently high sinus heart rate (HR) and/or an exaggerated HR response to minimal exertion, and can be responsible for palpitations, asthenia, chest pain, dizziness and syncope, which can be highly invalidating. Conventional treatment of IST, targeted to symptoms control, mainly consists on β-blockers. However, these drugs are often insufficient or not well tolerated because of side effects (mostly hypotension) that usually limit the administered dose. Ivabradine, a sinus rate lowering agent currently employed in Europe in the treatment of stable angina and chronic heart failure, has recently been demonstrated to be effective and safe in the treatment of IST by a few case reports and clinical trials. A randomized clinical trial comparing ivabradine to β-blockers has not be performed yet.

ELIGIBILITY:
Inclusion Criteria:

* Inappropriate sinus tachycardia (HR >100 bpm at rest ECG and/or medium Holter ECG HR >90 bpm)
* Age > 18 years;

Exclusion Criteria:

* Secondary causes of sinus tachycardia;
* Structural heart diseases,
* Postural orthostatic tachycardia syndrome;
* Sinus nodal reentrant tachycardia;
* Contraindications to beta-blockers;
* Administration of beta-blockers, non-di-hydropiridinic calcium channels antagonists, class I and III anti-arrhythmic drugs or digitalis at the time of enrollment;
* Age < 18 years;
* Inability of giving informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
heart rate reduction | three months
  Percentage of HR reduction at Holter ECG (mean, minimal and maximal)
heart rate reduction | three months
  Percentage of maximal HR reduction at stress-test ECG

SECONDARY OUTCOMES:
physical tolerance and quality of life | three months
  Improvement of stress-tolerance (maximal load reached at stress test ECG)
physical tolerance and quality of life | three months
  Improvement of the quality of life (Minnesota QoL questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Calò, FESC MD, Principal Investigator — Policlinico Casilino
Locations (1):
- Policlinico Casilino, Rome, Rome, Italy

REFERENCES:
- [Background] Calo L, Rebecchi M, Sette A, Martino A, de Ruvo E, Sciarra L, De Luca L, Zuccaro LM, Giunta G, Ciccaglioni A, Lioy E, Fedele F. Efficacy of ivabradine administration in patients affected by inappropriate sinus tachycardia. Heart Rhythm. 2010 Sep;7(9):1318-23. doi: 10.1016/j.hrthm.2010.05.034. Epub 2010 Jun 1. PMID 20621618
- [Background] Ptaszynski P, Kaczmarek K, Ruta J, Klingenheben T, Wranicz JK. Metoprolol succinate vs. ivabradine in the treatment of inappropriate sinus tachycardia in patients unresponsive to previous pharmacological therapy. Europace. 2013 Jan;15(1):116-21. doi: 10.1093/europace/eus204. Epub 2012 Jul 6. PMID 22772053